CLINICAL TRIAL: NCT02357667
Title: The Study of Cardiovascular Outcomes in Women With Preeclampsia Using Echocardiography: The SCOPE Study
Acronym: SCOPE
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa Levine, Clinical Instructor, Department of Obstetrics & Gynecology Division of Maternal Fetal Medicine, University of Pennsylvania
Other Study IDs: 821592
Record Dates: First submitted 2015-01-28; First posted 2015-02-06 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Evaluation of angiogenic factors, markers of heart failure, and evaluation of extracellular RNAs will specifically be used for discovery. The investigators will not be evaluating DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed cases: African American women with concern for severe preterm (37 weeks gestation) preeclampsia who are admitted to the inpatient obstetrical unit at HUP.
- Unexposed controls: African American women without preeclampsia or medical comorbidity who are matched by gestational age, maternal age, and BMI in the outpatient setting.

SUMMARY:
This study will evaluate the differences in cardiovascular parameters between women with severe preterm preeclampsia and those without preeclampsia using echocardiography and maternal blood. The investigators will also look at associations of abnormal cardiovascular findings and immediate complications among a high risk cohort of pregnant African American women.

DETAILED DESCRIPTION:
This will be a prospective cohort study. Exposed cases will be admitted to the inpatient obstetrical unit (labor & delivery or antepartum unit) at the Hospital of the University of Pennsylvania with concern for severe preterm preeclampsia. Unexposed controls will be matched by gestational age and other clinical factors and will be obtained from the outpatient setting (Helen O Dickens clinic or Penn ObGyn Associates at 3701 Market Street). The investigators will compare cardiovascular risk factors between these two groups.

ELIGIBILITY:
Exposed cases:

Inclusion Criteria:

* African American women who are admitted to the obstetrical unit with a concern for severe preeclampsia. Patients must be preterm (23-36 6/7 weeks) with a live singleton gestation and at least 18 years old. Women will baseline chronic hypertension and women on magnesium will be included.

Exclusion Criteria:

* Non-African American women, and African women with concern for severe preeclampsia who are admitted 23 weeks or 37 weeks. Women in labor will be excluded. Women with preexisting cardiovascular disease and women who are current smokers will be excluded.

Unexposed controls:

Inclusion Criteria:

* African American women obtaining prenatal care in our outpatient setting who meet matching criteria as noted above.

Exclusion Criteria:

* Non-African American women and women who are not receiving care at our institution.

  * All women who do not speak English and who are unable to be consented will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will take place on the obstetrical unit at the Hospital of the University of Pennsylvania (HUP) as well as in the outpatient setting. The patient population is primary from the surrounding urban region. The majority receive prenatal care at our institution. Based on fiscal year 2010 at HUP, the mean age was 24 years old and 85% were African American.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Cardiovascular parameters obtained on echocardiogram (longitudinal strain and E/E) | 2 years
Angiogenic factors and biomarkers of congestive heart failure (sFlt1) | 2 years

SECONDARY OUTCOMES:
Other cardiovascular parameters measured on echocardiogram (ventricular arterial coupling, arterial tonometry) | 2 years
Other angiogenic factors and biomarkers of CHF (VEGF, BNP, troponin, etc) | 2 years
Postpartum readmission rate | 2 years
Pulmonary edema during labor and delivery or postpartum | 2 years
Peripartum cardiomyopathy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, MD, Principal Investigator — UENN
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States